CLINICAL TRIAL: NCT01355146
Title: Non Interventional Study of Replagal® Home Therapy in Patients With Fabry Disease
Brief Title: Home Therapy With Replagal in Fabry Disease
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: Shire/CS02
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Fabry Disease
Keywords: Patients with proven Fabry's Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fabry's Disease under Replagal

SUMMARY:
The purpose of this study is to proof increasing patient satisfaction and preservation of quality of life in patients with Morbus Fabry disease receiving their Enzyme Replacement Therapy with Replagal (Agalsidase alfa) at home compared to receiving the infusions at the clinic or at doctor's practice.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female patient with a confirmed diagnosis of Fabry disease
* Age> 4 years
* Patient is under Replagal since at least 12 weeks ® therapy
* The patient is compliant, the previous Replagal ® infusions were performed approximately every 2 weeks in the center close to home or at the hospital / general practitioner at
* Patient has been well tolerated Replagal ® therapy, and there were in the last 12 weeks before inclusion in this study no significant infusion reactions to
* The patient has been selected before inclusion in this study for a home infusion therapy and has consented to (or their legal representative)
* The patient / be lawful. Representative has consented in writing to participate in this study.

Exclusion Criteria:

* Patient/legal representative does not give consent to participation in this study
* Patient/legal representative declines Replagal® home therapy
* The patient is participating in a clinical trial with a medicinal product

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with proven Fabry's Disease foreseen for home treatment with Agalsidase alfa at German Fabry centers
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2011-03-15 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction estimated on a 10-ary Likert scale | comparison of baseline to 12 months value

SECONDARY OUTCOMES:
Number (per infusion) and severity of infusion-related side effects | baseline compared to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (22):
- Austria (5):
  - Landeskrankenhaus Bregenz, Bregenz
  - LKH-Universitätsklinikum Graz, Graz
  - Paracelsus Medizinische Privatuniversität Salzburg, Salzburg
  - Universitätsklinik für Innere Medizin III, Vienna
  - Universitätsklinik für Kinder- und Jugendheilkunde, Vienna
- Germany (17):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinik II für Innere Medizin, Cologne
  - Med. Versorgungszentrum Dialyse-Centrum Cuxhaven, Cuxhaven
  - Alfried-Krupp-Krankenhaus Rüttenscheid, Essen
  - MVZ Immunologie am Krankenhaus Sachsenhausen, Frankfurt
  - Zentrum für Kinder und Jugendmedizin, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg, Giessen
  - Facharzt für Allgemeinmedizin, Hagen
  - Facharzt für Innere Medizin/Kardiologie, Höxter
  - Hans-Berger-Klinik für Neurologie, Jena
  - Universitätsklinikum Mainz, Zentrum für Kinder- und Jugendmedizin, Mainz
  - Private Practice, Dr. Glenn Sommer, Marienberg
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., München
  - Klinikum rechts der Isar, München
  - Landesklinikum St. Pölten, Neurologie, Pölten
  - Nephrologisches Zentrum Rendsburg, Rendsburg
  - Universitätsklinikum Ulm, Ulm

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fd24db2bf003ab46a7c